| Title | A Randomized Trial Assessing the Impact of |
|------------------|----------------------------------------------|
| | Educational Podcasts on Personal Control and |
| | Satisfaction During Childbirth |
| Short Title | LaPPS |
| NCT | NCT04933708 |
| Date of Document | 7/16/2021 |

#### **Labor Podcast Education for Patient Satisfaction**

#### What is involved in joining this research?

You will be approached during your pregnancy about the research project. At 28 weeks, you will be randomized to either receiving a link to podcasts that answer common questions about labor, or to usual patient education.

If you are randomized to receiving the link to podcasts, you may download and listen to the podcast on whatever app you choose and listen as many times as you'd like. You will also continue to receive the usual education about labor from your doctors and providers. If you are randomized to usual patient education, you will receive the usual education about labor from your doctors and providers.

After you deliver, you will receive a survey on your experience in labor as well as a postpartum depression screen via email or text (whichever you choose).

## What information about me may be collected, used or shared with others?

We will be collecting your name, telephone number or email address, and medical record number in order to follow you during your labor, birth, and postpartum period and send you the postpartum surveys. We will collect information regarding your labor and birth outcomes. This information will not be disclosed or shared with others outside of the researchers of this study.

### Why is my information being used?

Your information is used by the research team to contact you during the study. Your information and results of tests and procedures are used to:

- do the research
- oversee the research
- · to see if the research was done right
- to evaluate and manage research functions.

### Who may use and share information about me?

The following individuals may use or share your information for this research study:

- The investigator for the study and the study team:
  - o Dr. Sindhu Srinivas
  - o Dr. Fei Cai
- Other authorized personnel at Penn, including offices that support research operations
- Other research personnel with access to the databases for research and/or study coordination and as otherwise approved by the IRB

# Who, outside of the University of Pennsylvania, might receive my information?

#### Oversight organizations

• The U. S. Office of Human Research Protections (OHRP)

Once your personal health information is disclosed to others outside the School of Medicine, it may no longer be covered by federal privacy protection regulations.

The Principal Investigator or study staff will inform you if there are any additions to the list above during your active participation in the trial. Any additions will be subject to University of Pennsylvania procedures developed to protect your privacy.

# How long may the University of Pennsylvania use or disclose my personal health information?

Your authorization for use of your personal health information for this specific study will not expire.

Your information may be held in a research database. However, the School of Medicine may not re-use or re-disclose information collected in this study for a purpose other than this study unless:

- You have given written authorization
- The University of Pennsylvania's Institutional Review Board grants permission
- As permitted by law

# Can I change my mind about giving permission for use of my information?

Yes. You may withdraw or take away your permission to use and disclose your health information at any time. You do this by sending written notice to the investigator for the study. If you withdraw your permission, you will not be able to stay in this study.

## What if I decide not to give permission to use and give out my health information?

Then you will not be able to be in this research study.

You will be given a copy of this Research Subject HIPAA Authorization describing your confidentiality and privacy rights for this study.

By signing this document, you are permitting the School of Medicine to use and disclose personal health information collected about you for research purposes as described above.

| Signature: | Date: |
|------------|-------|
|------------|-------|